CLINICAL TRIAL: NCT01117727
Title: Sensorimotor Rhythm Brain-Computer Interface Switch to Operate Assistive Technology
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Performance of BCI switch insufficient in pilot testing.
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I0003 - AT SMR Switch Control; 5R21HD054697 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot Testing (Experimental)
  Interventions: Device: Brain Computer Interface Switch

INTERVENTIONS:
Device: Brain Computer Interface Switch — Subjects will wear an EEG cap for 1-2 hours typical per session and use the brain computer interface to operate assistive technology. Subjects will be asked to participate in 14-20 sessions.

SUMMARY:
The purpose of this research is to develop tools to help people who are paralyzed. These tools are called brain-computer interfaces (BCIs). BCIs would allow a person to use brain signals to operate technology. Specifically this project's goal is to design a BCI to operate a switch.

DETAILED DESCRIPTION:
The investigators want to make a BCI that can be used to operate commercially available technologies for communication, environmental control or computer access. The BCI would replace a switch to let people operate these technologies without moving. However, investigators need people to test the BCI so they can determine how effective it is in replacing a switch.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to read text on a computer screen
* Able to understand and remember instructions concerning participation

Exclusion Criteria:

* Unable to give informed consent
* Unable to understand and follow instructions
* Have abnormal tone or uncontrolled movements in the head-and-neck that would interfere with EEG recordings
* Known to have photosensitive epilepsy
* Open head lesions or sores

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Direct Brain Interface Project, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot Testing
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Testing
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Using the BCI as a Switch to Select From 4 Targets Using Scanning
Description: Average accuracy for selecting one of 4 targets with a switch operated by a brain-computer interface controlled by power in the sensorimotor rhythms. The 8 sessions were conducted over a 2 month period. Accuracy was calculated as the percentage of trials in which the target was correctly selected. Trials for all sessions were combined to create the overall average. Therefore, there is no standard deviation. .
Time Frame: 8 sessions over 2 months
Measure: Number; unit: percent of correct targets selected
Groups:
- Pilot Testing, 0.65 Scan Rate: Pilot subject testing protocol with scan rate at 0.65 seconds per item.
- Pilot Testing With Scan Rate at 2 Stdev: Pilot testing with scan rate set at twice the standard deviation of the reaction time.
Arm/Group | Pilot Testing, 0.65 Scan Rate | Pilot Testing With Scan Rate at 2 Stdev
Number analyzed (Participants) | 1 | 1
percent of correct targets selected | 60.5 | 78.4

ADVERSE EVENTS:
Arm/Group | Pilot Testing
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No